CLINICAL TRIAL: NCT03758300
Title: Radiofrequency Facilitates the Prehabilitation Process in Patients Undergoing Total Knee Arthroplasty: Effects on Preoperative and Postoperative Functional Capacity. A Double Blind Randomized Controlled Trial
Brief Title: RF TKA Prehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, JF Asenjo, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-3664
Record Dates: First submitted 2018-08-20; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency group (Experimental): In this group patients will receive in a sterile fashion continuous radiofrequency for 4 minutes to the 3 genicular nerves in the operative knee as well as Pulsed Radiofrequency at 42 degrees celsius, for 4 minutes (60-70 volts) to the saphenous nerve and the nerve to the Vastus Medialis, at the level of the adductor canal. The procedure is done under local anesthesia on an ambulatory basis. After the radiofrequency, Ropivacaine 0.5% 5 ml is injected to each one of the nerves, along with 5 milligrams of Methylprednisolone to each nerve. Once the procedure is completed (takes about 20 minutes), patients will be observed in the preoperative program facility for 30 minutes and then discharged home.
  Interventions: Other: Radiofrequency
- Control (Sham Radiofrequency) group (Sham Comparator): In this group patients will receive injections of the local anesthetic and steroids in the same anatomical locations, without activating the radiofrequency generator.
  Interventions: Other: Radiofrequency

INTERVENTIONS:
Other: Radiofrequency — See previous page

SUMMARY:
The purpose of this study is to compare the effects of the radiofrequency applied to the sensory innervation of the knee, with respect to a control group (standard therapy), in a prehabilitation program aiming to improve the functional recovery of patients undergoing TKA.

In the present study, the investigators hypothesize that participants treated with radiofrequency 4-6 weeks before the surgery, should be able to effectively accomplish the prehabilitation program and, therefore, have a faster recovery of their functional status in the post operative period , compared with the control group (That use the present state of the art approach)

DETAILED DESCRIPTION:
Postoperative functional capacity following TKA surgery has been strongly associated with preoperative functional status. Presence of pain, poor strength and flexibility, and limited ability to complete physiological tasks have been shown to be consistent predictors of poor recovery from knee surgery.

The postoperative period is associated with 30-40% decrease in functional capacity, and efforts have been made to facilitate the recovery by implementing rehabilitative measures over the period of weeks and months. However, the postoperative period might not be the best time to engage patients in intensive physiotherapy as they are easily tired and in pain. Preparing patients for the stress of surgery, called also prehabilitation, is emerging as a mean to optimize pre-operative status and increase functional reserve thus, increasing surgical stress tolerance. Observational and randomized controlled studies in patients scheduled for colorectal, thoracic, and spinal surgeries have suggested that a 4-6 weeks of moderate preoperative physical activity can lead to significant postoperative improvements in cardiorespiratory reserve and functional capacity. However, preliminary trials on the effect of a 6-8 weeks prehabilitation program with structured exercises prior to knee arthroplasty have reported contrasting results, and one of the reasons might be the high levels of pain encountered by these patients while exercising, therefore making it difficult to engage them in achieving effective prehabilitation. It would therefore, make sense if efforts were directed towards relieving pain thus, facilitating broader fitness enhancement strategies and improving the surgical experience and the recovery process.

Common pharmacological methods to relieve osteoarthritic pain while waiting for surgery, include acetaminophen, non-steroidal anti-inflammatory drugs (NSAIDS and Cox-2 inhibitors) and occasionally opioids. Non-surgical interventions, such as intra-articular injection with steroids or hyaluronic acids, acupuncture and periosteal stimulation therapy, are often used as complementary therapies of limited benefit. The use of pulsed and Continuous radiofrequency (PRF and CRF) to the saphenous nerve and the genicular nerves branches of the knee, have been shown to decrease significantly pain scores in 44% of patients with chronic OA of the knee for up to one year after the treatment. Akbasa et al. using the Western Ontario and McMaster Osteoarthritis Index (WOMAC), reported significant reduction of pain at rest, movement and flexion of the knee and increase in patient's satisfaction 6 months after the PRF treatment. Our group has recently demonstrated the benefits of radiofrequency treatment in patients waiting for total knee replacement TKA 9. More so, the investigators recent results reported to the American Society of Regional Anesthesia and Pain, showed in a randomized controlled trial promising results in terms of faster recovery of patients undergoing TKA, when they received RF instead of the standard postoperative analgesia technique 10.

The present study is, as mentioned above, related to an already approved and finished study in this institution: 15-209-MUHC "Functional outcome and postoperative analgesia following total knee arthroplasty: a prospective, randomized, double blind comparison between continuous adductor canal block and pulsed radiofrequency of saphenous and genicular nerves of the knee". In that study, our research group was investigating the effects of the Radiofrequency treatment preoperatively on the postoperative pain and functional recovery, in patients who did not participate in a prehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Chronic knee pain, with Dynamic VAS ≥ 5
* Scheduled for elective total knee arthroplasty
* Functional impairment due to pain because of knee osteoarthritis
* Taking medications to control the pain.
* Ability to perform the 6 MWT.

Exclusion Criteria:

* ASA physical status > 3
* Morbid obesity (BMI >40)
* Revision of total knee arthroplasty
* Mayor neuropsychiatric disease
* Mayor cardiac, renal or hepatic failure
* Anemia (hematocrit <30%)
* Immunosuppression
* Rheumatoid arthritis
* Allergy to opioids, to local anesthetics or other medications used in the study,
* Chronic regular use of large doses of opioids (>20mg equivalent of morphine/day) or sedatives
* Unwillingness to have spinal anesthesia
* History of recent drug abuse
* Contraindication to receive regional anesthesia (e.g. coagulation defect)
* Inability to walk before the surgery
* Inability to perform physical tasks
* Contraindications to physical exercise and training
* Prior mayor knee surgery
* Connective tissue diseases affecting the knee
* Serious neurologic disorders
* Injection with steroids or hyaluronic acids during the previous 3 months
* Active sciatic pain
* Anticoagulant medications

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
change of 15% of the total distance walked during a 6MWT | 18 weeks
  change of 15% or more in total distance in six minute walk test from baseline

SECONDARY OUTCOMES:
Change in WOMAC score | Baseline and 18 weeks
  Change in score of WOMAC questionnaire
Change in knee pain levels assessed by VAS (Dynamic/Static) | Baseline and 18 weeks
Change in amount of daily pain relief medication consumption | Baseline and 18 weeks
Change in total time of the time up and go (TUG) test | Baseline and 18 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided